CLINICAL TRIAL: NCT00985907
Title: Phase I/II Study of Liposomal Doxorubicin (Doxil®)/Melphalan/Bortezomib (Velcade®) in Relapsed/Refractory Multiple Myeloma
Brief Title: Doxil® + Melphalan + Velcade (DMV) in Relapsed/Refractory Multiple Myeloma
Acronym: DMV
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04262; NCI-2011-01238 (Registry Identifier: University of California, San Francisco)
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Multiple Myeloma; Patient Participation
Keywords: myeloma; DMV
MeSH Terms: conditions — Multiple Myeloma; Patient Participation; Neoplasms, Plasma Cell | interventions — liposomal doxorubicin; Melphalan; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doxil® + Melphalan + Velcade (DMV) (Experimental)
  Interventions: Drug: Doxil, melphalan, bortezomib

INTERVENTIONS:
Drug: Doxil, melphalan, bortezomib — Doxil®: IV over 30-60 min, Day 1 q28d
  Melphalan: IV over 30 min, Day 1 q28d
  Velcade®: IV bolus, Day 1, 4, 8, 11 q28d
  Dose Level 1: Doxil 10 mg/m2, Melphalan 5 mg/m2, Velcade 0.7 mg/m2
  Dose Level 2: Doxil 10 mg/m2, Melphalan 10 mg/m2, Velcade 0.7 mg/m2
  Dose Level 3: Doxil 20 mg/m2, Melphalan 10 mg/m2, Velcade 0.7 mg/m2
  Dose Level 4: Doxil 20 mg/m2, Melphalan 10 mg/m2, Velcade 1.0 mg/m2
  Other Names: Doxil, melphalan, Velcade

SUMMARY:
The median overall survival (OS) of relapsed/refractory multiple myeloma (MM) is less than nine months. However, phase II data with the proteasome inhibitor bortezomib (Velcade®) has been heartening, with 35% overall response rates and median survival of 16 months. In-vitro data has shown that this agent dramatically increases the sensitivity to chemotherapeutic agents. Liposomal doxorubicin (Doxil), melphalan, and bortezomib all have different mechanisms of action and toxicity profiles. Clinical studies employing two drug combinations with these agents in patients with refractory MM have found favorable efficacy (nearly no progression of disease) and tolerance data. Thus, the investigators are initiating a phase I/II study to examine the safety and efficacy of combining all three agents into the regimen DMV (Doxil® + melphalan + Velcade).

DETAILED DESCRIPTION:
Dose Level 1: Doxil 10 mg/m2, Melphalan 5 mg/m2, Velcade 0.7 mg/m2

Dose Level 2: Doxil 10 mg/m2, Melphalan 10 mg/m2, Velcade 0.7 mg/m2

Dose Level 3: Doxil 20 mg/m2, Melphalan 10 mg/m2, Velcade 0.7 mg/m2

Dose Level 4: Doxil 20 mg/m2, Melphalan 10 mg/m2, Velcade 1.0 mg/m2

Adjunctive therapy with a bisphosphonate, either pamidronate or zoledronic acid, will be given monthly.

Dose Escalation Schedule: Dose escalation will occur only after patients have completed at least two cycles at a given dose level.

1. If 0/3 experience DLT (as defined in attachment Section 6.0), the next three patients will be escalated by one dose level.
2. If 1/3 experience DLT, 3 additional patients enrolled at this dose level.

   * If 0, 1, or 2 of these additional patients experience DLT (i.e. total 3/6), the dose will be escalated.
   * If 3/3 experience DLT (i.e. total 4/6) then the next lower dose will be considered the MTD..
3. If 2/3 experience DLT, 3 additional patients enrolled at this dose level.

   * If 0 or 1 of these additional patients experience DLT (i.e. total 3/6), the dose will be escalated.
   * If 2 or more/3 experience DLT (i.e. total more than 3/6) then the next lower dose level is MTD

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics:

1. Patient previously diagnosed with multiple myeloma; Durie-Salmon Stage I, II, or III based on standard criteria
2. Progressive disease. For non-secretory multiple myeloma, progressive disease is defined as bone marrow biopsy with > 25% increase in plasma cells or an absolute increase of at least 10% over prior known level. Alternatively, development of new or worsening of existing lytic bone lesions or soft tissue plasmacytomas, or hypercalcemia (serum calcium >11.5 mg/dL), or relapse from complete response.

Patient Characteristics:

1. 18 yrs or older
2. Patient has given voluntary written informed consent.
3. Unless post-menopausal or surgically sterilized, a female must be willing to use an acceptable method of birth control
4. Male patient must agree to use an acceptable method for contraception for the duration of the study.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
6. Life expectancy is at least 3 months.
7. • Absolute Neutrophil Count (ANC) over 1,000/ul without the use of colony stimulating factors

   * Platelets over 50,000/ul without transfusion support 7 days
   * Bilirubin 2.0 mg/dl or less
   * aspartate aminotransferase (AST) 4 times or less upper limit normal Prior Therapy for Multiple Myeloma: Patients must have had at least 2 prior therapeutic regimens

Exclusion Criteria:

* Pregnant or breast feeding
* History of allergic reaction to compounds containing boron or mannitol.
* Active uncontrolled viral (including HIV), bacterial, or fungal infection.
* Grade III or IV toxicity due to previous anti-neoplastic therapy
* More than Grade 2 motor or sensory neuropathy
* Myocardial infarction within 6 months of enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled arrhythmias, or electrocardiographic evidence of acute ischemia.
* For any patients whose lifetime cumulative doxorubicin dose exceeds 400mg/m2, patients with left ventricular ejection fraction (LVEF) less than 35% by multigated acquisition (MUGA) .
* Concurrent administration of liposomal doxorubicin, melphalan, and bortezomib (single or two drug combinations of these are permissible)
* Less than 3 weeks since most recent chemotherapy or concurrent chemotherapy
* Use of corticosteroids (mroe than 10 mg prednisone/day or equivalent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2004-10-28 (Actual); Primary Completion 2008-10-07 (Actual); Study Completion 2010-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Martin, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - St. Vincent's Comprehensive Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Arms/Groups are not separated by individual cohorts within Phase 1 as information was lost when it was transferred from our legacy system. Paper records were lost in a flood, so participants were only grouped electronically by which phase they were enrolled. The study was terminated and participants were not enrolled in Phase 2 part of the study.
Groups:
- Phase 1: Doxil, melphalan, bortezomib: Doxil®: IV over 30-60 min, Day 1 q28d
  Melphalan: IV over 30 min, Day 1 q28d
  Velcade®: IV bolus, Day 1, 4, 8, 11 q28d
  Dose Level 1: Doxil 10 mg/m2, Melphalan 5 mg/m2, Velcade 0.7 mg/m2
  Dose Level 2: Doxil 10 mg/m2, Melphalan 10 mg/m2, Velcade 0.7 mg/m2
  Dose Level 3: Doxil 20 mg/m2, Melphalan 10 mg/m2, Velcade 0.7 mg/m2
  Dose Level 4: Doxil 20 mg/m2, Melphalan 10 mg/m2, Velcade 1.0 mg/m2
Period: Overall Study
Arm/Group | Phase 1
Started | 13
Completed | 0
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: Arms/Groups are not separated by individual cohorts within Phase 1 as the information was lost when it was transferred from our legacy system. Paper records were lost in a flood. So the participants were only grouped electronically by which phase they were enrolled
Arm/Group | Doxil® + Melphalan + Velcade (DMV)
Number analyzed (Participants) | 13
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1
  40-49 years old | 1
  50-59 years old | 6
  60-69 years old | 3
  70-79 years old | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT) (Phase 1)
Description: Safety assessments will be evaluated as the proportion of patients experiencing the following: treatment-related grade 3 or higher toxicity (hematologic and nonhematologic) and treatment-related death.
Time Frame: Up to 2 cycles of treatment, approximately 56 days
Population: Only data for Phase 1, Cohort 1 DLT was collected
Measure: Count of Participants; unit: Participants
Arm/Group | Doxil® + Melphalan + Velcade (DMV)
Number analyzed (Participants) | 4
Participants | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase 1)
Description: The MTD will be considered the dose below where <= 3 patients experience a DLT and the dose that two cycles can be given without meeting toxicity criteria.
Time Frame: Up to 1 year
Population: Data not collected
Arm/Group | Doxil® + Melphalan + Velcade (DMV)
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of All Treatment-related Toxicities at the MTD (Phase 1)
Description: NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3 will be used to determine all treatment related toxicities at the MTD. Participants entered at the MTD Dose level from the phase I portion of the study will also be included in this analysis
Time Frame: 5 years
Population: Data not collected
Arm/Group | Doxil® + Melphalan + Velcade (DMV)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Response Rate
Description: At each cycle, participants will be assessed for treatment response: Complete Response (CR), Near CR(nCR), Partial Response (PR), Minimal Response (MR), Stable Disease (SD), or Progressive Disease (PD) on at least 2 measurements at minimum of a 4 week interval. The overall response rate will use the best response of CR, nCR, PR, MR, or SD. In order to qualify for responses, the following events may NOT have occurred - new/increased size of plasmacytomas or bone lesions, recurrence or persistence of hypercalcemia. Collapse of bony structure from previous disease will not constitute progression or failure to respond. Participants entered at the MTD Dose level from the phase I portion of the study will also be included in this analysis
Time Frame: Up to 5 years
Population: Data not collected
Arm/Group | Doxil® + Melphalan + Velcade (DMV)
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Response (Phase 2)
Description: Efficacy of DMV as determined by time to first observed response. Participants entered at the MTD Dose level from the phase I portion of the study will also be included in this analysis
Time Frame: 28 days
Population: Data not collected
Arm/Group | Doxil® + Melphalan + Velcade (DMV)
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression-free Survival (Phase 2)
Description: Efficacy of DMV as determined by progression free survival. Participants entered at the MTD Dose level from the phase I portion of the study will also be included in this analysis
Time Frame: Up to 5 years
Population: Data not collected
Arm/Group | Doxil® + Melphalan + Velcade (DMV)
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Survival (Phase 2)
Description: Overall survival is defined as the amount of time from start of study therapy until death, or study completion. Participants entered at the MTD Dose level from the phase I portion of the study will also be included in this analysis
Time Frame: Up to 5 years
Population: Data not collected
Arm/Group | Doxil® + Melphalan + Velcade (DMV)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Arms are not separated by individual cohorts within Phase 1 as information was lost when it was transferred from legacy system. When legacy patient data was transferred, it was decided that only mortality and serious adverse event data should be retained and transferred. Other adverse event (AE) data was not electronically transferred. Paper records were lost in a flood, so participants AE data could not be recovered. The study was terminated and participants not enrolled in Phase 2.
Groups:
- Phase 1 Doxil® + Melphalan + Velcade (DMV): Doxil, melphalan, bortezomib: Doxil®: IV over 30-60 min, Day 1 q28d
  Melphalan: IV over 30 min, Day 1 q28d
  Velcade®: IV bolus, Day 1, 4, 8, 11 q28d
  Dose Level 1: Doxil 10 mg/m2, Melphalan 5 mg/m2, Velcade 0.7 mg/m2
  Dose Level 2: Doxil 10 mg/m2, Melphalan 10 mg/m2, Velcade 0.7 mg/m2
  Dose Level 3: Doxil 20 mg/m2, Melphalan 10 mg/m2, Velcade 0.7 mg/m2
  Dose Level 4: Doxil 20 mg/m2, Melphalan 10 mg/m2, Velcade 1.0 mg/m2
Arm/Group | Phase 1 Doxil® + Melphalan + Velcade (DMV)
All-Cause Mortality (participants affected / at risk) | 2/13
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Doxil® + Melphalan + Velcade (DMV) (N=13)
Hyperbilirubinemia (Investigations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was terminated early due to low accrual in Phase 1. No participants were enrolled in Phase 2. Participant flow, baseline, and adverse event data was electronically transferred from a legacy clinical trials database by phase group only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No